CLINICAL TRIAL: NCT01095120
Title: A Phase II Study of Tesetaxel Administered at a Flat Dose Once Every 21 Days as Second-line Therapy to Subjects With Advanced Gastric Cancer
Brief Title: Tesetaxel as Second-line Therapy for Patients With Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Genta Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOG201
Record Dates: First submitted 2010-03-26; First posted 2010-03-29 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Adenocarcinoma of the Stomach; Adenocarcinoma of Esophagogastric Junction
MeSH Terms: interventions — tesetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Tesetaxel — For subjects in Cohort A, a flat dose of 40 mg will be administered in Cycle 1; the dose will be adjusted based on body weight. In subsequent cycles, depending on tolerability, the Cycle 1 flat dose may be increased by 5 mg in Cycle 2, and the Cycle 2 flat dose may again be increased by 5 mg in Cycle 3.
  For subjects in Cohort B, a flat dose of 50 mg will be administered in Cycle 1; the dose will be adjusted based on body weight. In subsequent cycles, depending on tolerability, the dose may be increased by 10 mg in Cycle 2.
  For subjects in Cohort C, a dose of 27 mg/m2 will be administered in Cycle 1. In subsequent cycles, depending on tolerability, the dose will be increased to 35 mg/m2 in Cycle 2.
  Other Names: DJ-927

SUMMARY:
Tesetaxel is an orally administered chemotherapy agent of the taxane class. This study is being undertaken to evaluate the efficacy and safety of tesetaxel administered as second-line therapy to patients with advanced gastric cancer.

ELIGIBILITY:
Primary inclusion criteria:

* Confirmed diagnosis of adenocarcinoma of the stomach or esophagogastric junction
* Measurable disease (revised RECIST; Version 1.1) based on computed tomography
* Eastern Cooperative Oncology Group performance status 0 or 1
* Treatment with only 1 prior regimen (as first-line therapy) and that regimen included a fluoropyrimidine and/or a platinum analogue
* Documented disease progression within 4 months of the last dose of the 1 prior regimen
* Adequate bone marrow, hepatic, and renal function, as defined in the protocol
* At least 4 weeks and recovery from effects of prior surgery or other therapy, including immunotherapy, radiation therapy, or cytokine, biologic or vaccine therapy, with an approved or investigational agent
* Ability to swallow an oral solid-dosage form of medication

Primary exclusion criteria:

* Nonmeasurable disease only (revised RECIST; Version 1.1)
* History or presence of brain metastasis or leptomeningeal disease
* Operable gastric cancer or operable cancer of the esophagogastric junction
* Uncontrolled diarrhea, defined as more than 3 loose bowel movements above the patient's usual number of bowel movements on at least 2 days within the 14 days prior to enrollment
* Uncontrolled nausea or vomiting within the 14 days prior to enrollment despite the administration of standard antiemetic therapy
* Known malabsorptive disorder
* Significant medical disease other than cancer, as defined in the protocol
* Presence of neuropathy > Grade 1 (National Cancer Institute Common Toxicity Criteria [NCI CTC]; Version 4.0)
* Prior treatment with a taxane or other tubulin-targeted agent (eg, indibulin) other than a vinca alkaloid
* Need to continue any regularly-taken medication that is a potent inhibitor or inducer of the CYP3A pathway or P-glycoprotein activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-09 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Response rate (Response Evaluation Criteria In Solid Tumors (RECIST)) | 12 months from date of first dose of study medication

SECONDARY OUTCOMES:
Disease control rate (ie, the percentage of patients with a confirmed complete or partial response [of any duration] or stable disease at least 6 weeks in duration) | 12 months from date of first dose of study medication
Durable response rate (ie, the proportion of patients with a confirmed complete or partial response at least 6 months in duration) | 12 months from date of first dose of study medication
Duration of response | 12 months from date of first dose of study medication
Adverse events | Through 30 days post last dose of study medication

CONTACTS AND LOCATIONS:
Overall Officials: Jaffer Ajani, MD, Study Chair — M.D. Anderson Cancer Center
Locations (4):
- United States (3):
  - Northwestern Medical Faculty Foundation, Chicago, Illinois
  - Abramson Cancer of the University of Pennsylvania at Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - The University of Texax MD Anderson Cancer Center, Houston, Texas
- Severance Hospital, Yonsei University Health System, Seoul, South Korea